CLINICAL TRIAL: NCT05710978
Title: Biomarkers to Assess Acute Kidney Injury Risk During Heat Strain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Grant proposal was not funded
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Riana Pryor, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STUDY00005847-Pilot
Record Dates: First submitted 2023-01-18; First posted 2023-02-02 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Hyperthermia; Kidney Injury, Acute
MeSH Terms: conditions — Hyperthermia; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Work Heat Stress (Experimental): Each participant will complete three consecutive days of heavy intensity aerobic work in a hot environment.
  Interventions: Other: Work Protocol

INTERVENTIONS:
Other: Work Protocol — Participants will complete 4 hours of walking and cycling to a work:rest ratio of 3:1.

SUMMARY:
Prolonged, high intensity work in a hot environment results in significant strain on the body, known as heat strain. Heat strain in hot occupational settings such as agriculture, fire suppression, and military work can lead to ~20% of workers exceeding the glomerular filtration rate indicated thresholds for acute kidney injury (AKI). However, it is unclear whether these individuals truly experienced AKI or if these were normal, healthy physiologic responses. To better determine if AKI occurs in the staggering number of workers previously reported, AKI biomarkers are needed in addition to kidney function markers (e.g., glomerular filtration rate) to characterize this response. The product of urinary tissue inhibitor of metalloproteinase 2 (TIMP-2) and insulin-like growth factor binding protein 7 (IGFBP7) is a promising Food and Drug Administration approved biomarker indicating risk of AKI and is currently used in hospitalized individuals. The usefulness of this biomarker in determining AKI in healthy individuals during heat strain is now beginning to be understood. Consecutive days of heat strain can result in repeated AKI, which is hypothesized to lead to chronic kidney disease. There is an epidemic of chronic kidney disease of non-traditional causes occurring in workers who undergo repeated days heat strain, including approximately 15% of outdoor workers in Central America. Of the few studies that investigated consecutive days of work in the heat, we demonstrated that participants exceed the glomerular filtration rate indicated threshold for AKI during consecutive days of heat strain. This project will determine whether [TIMP-2 x IGFBP7] increases during occupational relevant heat exposures in a healthy, active population. Additionally, this project will compare the impact of repeated exposures to a hot environment on risk of AKI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals (18-39 years old)
* Regularly completes aerobic exercise at least 60 min per week

Exclusion Criteria:

* History of cardiovascular, metabolic, respiratory, neural, or renal disease
* Hypertensive or tachycardic during the screening visit (systolic blood pressure > 139 mmHg, diastolic blood pressure > 89 mmHg, heart rate > 100 bpm)
* Current tobacco or nicotine use or previous regular use within the past 2 years
* Current or previous musculoskeletal injury limiting physical activity
* Taking medications with known thermoregulatory or cardiovascular effects (e.g., aspirin, beta blockers, diuretics, psychotropics, etc.)
* A positive pregnancy test at any point during the study or currently breastfeeding
* Study physician discretion based on any other medical condition or medication

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
[TIMP-2 x IGFBP-7] concentration | Minute 0
  The product of [Tissue inhibitor of metalloproteinase 2 (TIMP-2) and Insulin-like growth factor binding protein 7 (IGFBP7)] is a biomarker that has the potential for prediction of acute kidney injury.
[TIMP-2 x IGFBP-7] concentration | Hour 4
  The product of [Tissue inhibitor of metalloproteinase 2 (TIMP-2) and Insulin-like growth factor binding protein 7 (IGFBP7)] is a biomarker that has the potential for prediction of acute kidney injury.
[TIMP-2 x IGFBP-7] concentration | Hour 5
  The product of [Tissue inhibitor of metalloproteinase 2 (TIMP-2) and Insulin-like growth factor binding protein 7 (IGFBP7)] is a biomarker that has the potential for prediction of acute kidney injury.

SECONDARY OUTCOMES:
NGAL concentration | Minute 0
  Neutrophil gelatinase-associated lipocalin (NGAL) measures kidney injury.
NGAL concentration | Hour 4
  Neutrophil gelatinase-associated lipocalin (NGAL) measures kidney injury.
NGAL concentration | Hour 5
  Neutrophil gelatinase-associated lipocalin (NGAL) measures kidney injury.
Serum creatinine concentration | Minute 0
  Serum creatinine concentration is a measure of kidney function.
Serum creatinine concentration | Hour 4
  Serum creatinine concentration is a measure of kidney function.
Serum creatinine concentration | Hour 5
  Serum creatinine concentration is a measure of kidney function.
Urine creatinine concentration | Minute 0
  Urine creatinine concentration is a measure of kidney function.
Urine creatinine concentration | Hour 4
  Urine creatinine concentration is a measure of kidney function.
Urine creatinine concentration | Hour 5
  Urine creatinine concentration is a measure of kidney function.

CONTACTS AND LOCATIONS:
Overall Officials: Riana R Pryor, PhD, Principal Investigator — University at Buffalo
Locations (1):
- Center for Research and Education in Special Environments, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No
Once published, pooled and de-identified data will be made available to interested researchers upon request.